CLINICAL TRIAL: NCT01263535
Title: Circadian Continuous Intraocular Pressure Monitoring With SENSIMED Triggerfish® Ocular Telemetry Sensor in Patients on Tafluprost Treatment
Brief Title: Use of an Ocular Telemetry Sensor in Tafluprost Treated Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Sensimed AG (Industry)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Dr Tarek Shaarawy, University Hospital Geneva
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09/06
Record Dates: First submitted 2010-12-02; First posted 2010-12-20 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-08

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SENSIMED Triggerfish (Experimental)
  Interventions: Device: SENSIMED Triggerfish

INTERVENTIONS:
Device: SENSIMED Triggerfish — Contact lens-based device for the continuous recording of IOP fluctuations, with a portable recording system

SUMMARY:
This clinical trial is designed to investigate the performance of SENSIMED Triggerfish® during 24-hour continuous IOP fluctuation monitoring, defined as the number of valid recording intervals over the 24-hour period.

The investigation will recruit male and female patients older than 18 years and diagnosed with glaucoma and treated with tafluprost in both eyes. 20 subjects will be enrolled in the study. Patients will be considered enrolled in the study upon signature of informed consent. A screening visit and one 24-hour IOP fluctuation monitoring session during a 36-hour hospitalisation, are planned for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years.
* Untreated IOP of ≥22 mmHg in both eyes.
* Documented, typical glaucomatous visual field (VF) loss (nasal step, or arcuate, paracentral or Seidel's scotoma) determined by automated static threshold perimetry (Octopus 100), and glaucomatous optic nerve head cupping (neural rim notching or saucerization) in both eyes.
* Patients under tafluprost treatment since at least 4 weeks in both eyes.
* Patients who accept signing an informed consent approved by the Ethics Committee.

Exclusion Criteria:

* Patients not able to understand the nature of the research
* Patients under tutorship
* Corneal abnormalities in both eyes
* Subjects with contraindications for wearing contact lenses
* History of ocular surgery within the last 3 months
* Known hypersensitivity to tafluprost or to any of its excipients
* Full-frame metal glasses during monitoring with SENSIMED Triggerfish®
* Pregnancy and lactation
* Simultaneous participation in other clinical research
* Patients with evidence of ocular infection or inflammation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-09; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Acquisition of 24-hour Sensor output signal | After 24-hour continuous recording
  Performance is assessed as the portion of valid data (actual number of valid data points recorded compared to expected number of recorded data points) during 24-hour recording.

SECONDARY OUTCOMES:
Possible IOP fluctuation | After 24-hour recording with study device
  Fluctuation is defined as a change of 25% or more from the mean Sensor output over 24 hours for each participant.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Geneva, Geneva, Switzerland